CLINICAL TRIAL: NCT03814954
Title: Nebulized Epinephrine Versus Nebulized Salbutamol in Bronchiolitis Among Children Aged 1month-24months
Brief Title: Nebulized Epinephrine vs. Salbutamol in Bronchiolitis Among Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Makassed General Hospital (Other)
Responsible Party: Principal Investigator, Mariam Rajab, Clinical professor, Makassed General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1812182
Record Dates: First submitted 2019-01-21; First posted 2019-01-24 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-08

CONDITIONS: Respiratory Distress Score
MeSH Terms: interventions — Albuterol; Epinephrine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Salbutamol (Active Comparator): Patients will receive salbutamol (2 units/kg) with 3 ml normal saline by nebulizer.
  Interventions: Drug: Salbutamol
- Epinephrine (Experimental): Patients will receive epinephrine (0.5 mg/dose) with 3 ml normal saline by nebulizer.
  Interventions: Drug: Epinephrine

INTERVENTIONS:
Drug: Salbutamol — At first day of admission, patients will receive 3 doses of nebulized salbutamol every 20 minutes. Then after 24 hours patients will receive standing dose according to clinical status
  Arms: Salbutamol
Drug: Epinephrine — At first day of admission, patients will receive 3 doses of nebulized epinephrine every 20 minutes. Then after 24 hours patients will receive standing dose according to clinical status
  Arms: Epinephrine

SUMMARY:
Acute bronchiolitis, mostly secondary to infection due to Respiratory syncytial virus (RSV) is very common in infants under two years old. It is usually benign. However, the dyspnea it causes is a big concern for parents and this disease can take a severe form on certain particular ground thus constituting a frequent reason for hospitalization in pediatrics. Nebulized epinephrine showed more efficacy than nebulized salbutamol.

DETAILED DESCRIPTION:
The objective of this study is to determine if nebulized epinephrine is more efficacious than nebulized salbutamol in all hospitalized children (1 month to 24 months) in treatment of bronchiolitis. A randomized clinical trial which recruits children admitted to the pediatrics department with diagnosis of bronchiolitis. Children aged 1 month to 2 years will be included in the study.

Children who meet the inclusion criteria will be alternately distributed in two groups:

Group 1:

Will receive salbutamol (2 units/kg) with 3 ml normal saline by nebulizer.

Group 2:

Will receive epinephrine (0.5 mg/dose) with 3 ml normal saline by nebulizer. All admitted patients will receive aerosol every 20 minutes three times and after, depending on the clinical status of the patients, they will be given oxygen therapy at 1.5 liters / minute at the admission if oxygen saturation is below 94% till the normalization of the oxygen saturation.

Clinical parameters such as clinical score, oxygen saturation with pulse oximetry, heart rate, and temperature will be measured at admission, at hour 1 to hour 12 and then every 24 hours until they are discharged.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with acute bronchiolitis.

Exclusion Criteria:

* Children with congenital heart disease or
* chronic lung diseases

Ages: 1 Month to 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Length of stay | 5 days
  Patients hospitalization duration will be recorded

SECONDARY OUTCOMES:
Respiratory distress scoring | 5 days
  The score will be measured through Silverman-Andersen Retraction scoring. The minimum score is 0 indicating no distress. The maximum score is 10 indicating severe respiratory distress

CONTACTS AND LOCATIONS:
Overall Officials: Mariam Rajab, MD, Principal Investigator — Makassed General Hospital
Locations (1):
- Makassed General Hospital, Beirut, Lebanon